CLINICAL TRIAL: NCT03435458
Title: Balloon to Induce Labor in Generous Women
Acronym: BIGW
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: interim analyses
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RC31/16/8911
Record Dates: First submitted 2018-02-09; First posted 2018-02-19 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Maternal Obesity
Keywords: Induced labor; Maternal obesity
MeSH Terms: conditions — Pregnancy in Obesity | interventions — Misoprostol

STUDY DESIGN:
Intervention Model Description: The study is a randomized, multicentre, open-label, controlled trial comparing association of balloon catheter plus oral prostaglandin E1 versus oral prostaglandin E1 alone to induce labor in a 1:1 randomization of nulliparous obese women.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balloon catheter + oral misoprostol (Experimental)
  Interventions: Combination Product: Balloon catheter + oral misoprostol
- Oral misoprostol alone (Active Comparator)
  Interventions: Drug: Oral misoprostol alone

INTERVENTIONS:
Combination Product: Balloon catheter + oral misoprostol — The pharmacological cervical ripening will be administered just after the balloon catheter insertion (after coming back in her room) and will consist of misoprostol 25 micrograms given orally (oral prostaglandin E1). The same dose will be given every 2 hours until beginning of labor with a maximum of 8 administrations.
  Arms: Balloon catheter + oral misoprostol
Drug: Oral misoprostol alone — Patients will receive a pharmacological cervical ripening alone that consist of Misoprostol 25 micrograms given orally (oral prostaglandin E1). The same dose will be given every 2 hours until beginning of labor with a maximum of 8 administrations.
  Arms: Oral misoprostol alone

SUMMARY:
The rate of obesity increases continuously in France as in many developing countries.The risk of cesarean delivery is increased in obese compared to normal-weight women and postpartum complications as infections, thromboembolic events and related maternal death, are more common among obese women who deliver by cesarean than both normal-weight women with caesarean deliveries and obese women with vaginal deliveries. Unfortunately, obesity is associated with a higher rate of failed induction requiring a cesarean delivery and especially in nulliparous.

Methods of induction for obese women have to be improved to decrease the c-section rate but investigators should also be cautious on the type and dose of PG not to affect the neonatal wellbeing associated with uterine hyperstimulation.

The aim of this study is to demonstrate the efficacy of the association of mechanical and pharmacological cervical ripening (balloon catheter plus 50 µg oral prostaglandin E1) versus pharmacological cervical ripening alone (50 µg oral prostaglandin E1) to reduce the rate of caesarean sections in nulliparous obese women.

DETAILED DESCRIPTION:
The rate of obesity increases continuously in France as in many developing countries. In 2012, in the US, one third of all pregnant women were obese. The risk of cesarean delivery is increased in obese compared to normal-weight women and postpartum complications as infections, thromboembolic events and related maternal death, are more common among obese women who deliver by cesarean than both normal-weight women with caesarean deliveries and obese women with vaginal deliveries.

Prevalence of post-term is increased in obese pregnant women and the rate of induction of labor is twice the rate of normal-weight women, 42% versus 23% in the 2010 French National Survey.

Unfortunately, obesity is associated with a higher rate of failed induction requiring a cesarean delivery and especially in nulliparous.

Methods of induction for obese women have to be improved to decrease the c-section rate but investigators should also be cautious on the type and dose of PG not to affect the neonatal wellbeing associated with uterine hyperstimulation.

In a recent randomized clinical trial (RCT), the rate of c-section after labor induction in obese women was not increased in obese women compared to normal-weight women with balloon catheter but it was also increased with prostaglandin E2 (PGE2) and moreover with higher rate of uterine hyperstimulation. Recently, low dose of oral misoprostol (PGE1) has been showed to be the drug with the lowest rate of c-section after induction of labor in all women and balloon catheter to be associated with the lowest rate of hyperstimulation. Because safety of these two specific methods for induction of labor, a comparison 1 to 1 were done recently for induction of labor in singletons with comparable results.

Very few studies have focused on induction of labor in obese women even if the rate of maternal and neonatal complications are higher.

The efficacy of combining these two methods with different mechanism of induction have been showed recently but no study has been published today on obese women. Recently a trial have showed a shorter induction-delivery time with the combination (misoprostol-foley) for induction of labor in the whole population with less need of oxytocin during labor without more complications neither for the mother nor for the baby.An induction will be considered "failed" if at least 12 hours have elapsed since both rupture of membranes and use of a uterine stimulant and the patient remains in latent labor.

The aim of this study is to demonstrate the efficacy of the association of mechanical and pharmacological cervical ripening (balloon catheter plus 50 µg oral prostaglandin E1) versus pharmacological cervical ripening alone (50 µg oral prostaglandin E1) to reduce the rate of caesarean sections in nulliparous obese women.

ELIGIBILITY:
Inclusion Criteria:

* female
* pregestational BMI ≥ 30 kg/m2 (weight/height2)
* singleton pregnancy with cephalic presentation
* nulliparous
* ≥ 36 weeks gestational age
* decision of induction of labor
* bishop score ≤ 5
* ≤ 3 uterine contractions / 10 min
* ≥ 18 years of age
* personally signed and dated informed consent document
* ability to comply with the requirement of the study
* insurance coverage

Exclusion Criteria:

* deceleration on Fetal Heart Rate (FHR)
* placenta praevia
* bleeding
* premature rupture of membrane
* chorioamnionitis
* allergy to prostaglandins
* contraindication to ballon
* active genital herpes infection
* HIV infection
* fetal serious congenital anomaly
* patient subject to a legal protection order

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 429 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Efficacy of the association of mechanical and low dose oral misoprostol compared to oral misoprostol alone, to reduce the rate of caesarean section of all indications in obese women. | Day 0 to day 2
  Assessed by the caesarean section occurrence whatever the indication (binary endpoint).

SECONDARY OUTCOMES:
Effectiveness criteria. | Day 0 to day 2
  Effectiveness criteria chosen for the cost-effectiveness analysis will be the caesarean section rate for all indications.
Cost analysis. | Day 0 to day 2
  Cost estimates, for the construction of ICER, will be performed from the health insurance perspective.
  Costs taken into account will be those related to the management of obese pregnant women during inpatient stays for the delivery in both arms (i.e. combining method vs. oral prostaglandin alone). They include the costs of initial hospitalization for delivery. The expenses incurred in the management of patients in each arm will be recorded over a the study follow-up.
Resources consumption collection. | Day 0 to day 2
  Resource consumption will be gathered prospectively in each arm, during the follow-up period using a bottom-up approach. Data will be collected from the Medical Information Departments of each center participating in the study for hospitalization costs.
Costs valuation. | Day 0 to day 2
  Hospital stays will be valued from the French framework of pricing, the hospital Activity "Tarification à l'activité" (T2A). Hospital stays linked to the patient's care in each strategy will be valued from the French Diagnosis Related Group (DRGs).
Cost-effectiveness analysis. | Day 0 to day 2
  A cost-effectiveness analysis will be performed from the health insurance perspective. An Incremental Cost Effectiveness Ratio (ICER) will be calculate to establish a link between costs and medical consequences, expressed in terms of rate of caesarian section rate, between the two strategies for labor induction.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Vayssiere, Pr, Principal Investigator — University Hospital, Toulouse
Locations (18):
- France (17):
  - CHU Clermont-Ferrand, Clermont-Ferrand, Auvergne-Rhône-Alpes
  - CHU St Etienne, Saint-Etienne, Auvergne-Rhône-Alpes
  - CHU Tours, Tours, Centre-Val de Loire
  - CHRU Lille, Lille, Hauts-de-France
  - CHU Saint Denis de la Reunion, Saint-Denis, La Réunion
  - CHU St Pierre de la Reunion, Saint-Pierre, La Réunion
  - CHU de Toulouse, Toulouse, Midi-Pyrénées
  - CHU Bordeaux, Bordeaux, Nouvelle-Aquitaine
  - CHU Nimes, Nîmes, Occitanie
  - Hôpital St Joseph, Marseille, Provence-Alpes-Côte d'Azur Region
  - CHU Montpellier, Montpellier
  - CHU Nantes, Nantes
  - CHU Poitiers, Poitiers
  - CHU Antoine Beclère, Clamart, Île-de-France Region
  - CHU Kremlin Bicêtre, Le Kremlin-Bicêtre, Île-de-France Region
  - Centre hospitalier St Joseph, Paris, Île-de-France Region
  - CHI Poissy, Poissy, Île-de-France Region
- CHU Fort de France, Fort-de-France, Martinique

REFERENCES:
- [Background] Battarbee AN, Palatnik A, Peress DA, Grobman WA. Association of Early Amniotomy After Foley Balloon Catheter Ripening and Duration of Nulliparous Labor Induction. Obstet Gynecol. 2016 Sep;128(3):592-597. doi: 10.1097/AOG.0000000000001563. PMID 27500341
- [Background] Connolly KA, Kohari KS, Rekawek P, Smilen BS, Miller MR, Moshier E, Factor SH, Stone JL, Bianco AT. A randomized trial of Foley balloon induction of labor trial in nulliparas (FIAT-N). Am J Obstet Gynecol. 2016 Sep;215(3):392.e1-6. doi: 10.1016/j.ajog.2016.03.034. Epub 2016 Mar 24. PMID 27018464
- [Background] McMaster K, Sanchez-Ramos L, Kaunitz AM. Evaluation of a Transcervical Foley Catheter as a Source of Infection: A Systematic Review and Meta-analysis. Obstet Gynecol. 2015 Sep;126(3):539-551. doi: 10.1097/AOG.0000000000001002. PMID 26244535
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264